CLINICAL TRIAL: NCT03961984
Title: Long-term Follow-up of Anal Fistula Plug for Treatment of Complex Trans-sphincteric Fistulas
Brief Title: Long-term Follow-up of Anal Fistula Plug
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: Plug follow-up 2006
Record Dates: First submitted 2019-05-08; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Anal Fistula
Keywords: anal fistula; fistula-in-ano; surgical plug; collagen plug; complex anal fistula; transsphincteric anal fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Punctal Plugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Complex anal fistula: Patients with complex transsphincteric anal fistulas were treated with Biodesign® plug.
  Interventions: Procedure: Biodesign® anal fistula plug

INTERVENTIONS:
Procedure: Biodesign® anal fistula plug — Patient in general anesthesia and lithotomy position. Mucosa excision of the internal fistula opening is performed. The plug was prepared in 0.9% sodium chloride, and secured to the endoluminal brush by a suture with a 2-0 vicryl tie. The narrow end of the of the plug was then pulled through the internal opening into the fistula tract. The plug was pulled until it covered the whole length of the fistula and blocked the internal opening, the excess plug material coming out through the external opening. The plug was fixed at the internal opening by reabsorbable 3-0 sutures. Special attention was paid to ensuring that the plug was covered by mucosa when closing the internal opening. The excess plug material was trimmed by the external opening that was left open for drainage.
  Other Names: Surgisis anal fistula plug; Collagen plug

SUMMARY:
Aim of the study is to evaluate long-term success rate of Biodesign® anal fistula plug for treatment of complex trans-sphincteric anal fistulas.

DETAILED DESCRIPTION:
A prospective series of 95 consecutive patients (30 with inflammatory bowel disease) treated with Biodesign® plug in May 2006 - October 2009. All patients were preoperatively assessed by physical examination and 3D endoanal ultrasound, and treated with a loose seton. The patients were assessed by physical examination and 3D endoanal ultrasound at 2 weeks, 3 months, and 6 to 12 months after surgery. Long-term follow-up was carried out using a questionnaire, and, when indicated, physical examination and 3D endoanal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* complex transsphincteric anal fistula

Exclusion Criteria:

* ano/rectovaginal fistula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with anal fistulas not treatable with a simple fistulotomy offered to participate.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Fistula recurrence; Technical failure | Week 2
  Plug fallen out
Fistula recurrence; Infection | Week 2
  Surgical site infection
Fistula recurrence; Infection | Month 3
  Surgical site infection
Fistula recurrence; Infection | Month 6-12
  Surgical site infection
Fistula recurrence; Infection | Through study completion, an average of 8 years
  Surgical site infection
Fistula recurrence; New opening | Week 2
  Faeces coming through external opening
Fistula recurrence; New opening | Month 3
  Faeces coming through external opening
Fistula recurrence; New opening | Month 6-12
  Faeces coming through external opening
Fistula recurrence; New opening | Through study completion, an average of 8 years
  Faeces coming through external opening

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Starck, MD, PhD, Study Chair — Region Skane
Locations (1):
- Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Aho Falt U, Zawadzki A, Starck M, Bohe M, Regner S, Johnson LB. Postoperative three-dimensional endoanal ultrasound findings and relation to anal fistula plug failure. Scand J Gastroenterol. 2023 Jul-Dec;58(10):1200-1206. doi: 10.1080/00365521.2023.2212310. Epub 2023 May 18. PMID 37203207